CLINICAL TRIAL: NCT02674633
Title: A Randomized, Controlled, Parallel-group, Intervention Study to Assess At-home, Game-based Digital Therapy for Treating Pediatric Participants Ages 8 to 12 Years Old With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Software Treatment for Actively Reducing Severity of ADHD
Acronym: STARS-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Akili-001R
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Minimum number of subjects = 300, Anticipated number of subjects = 330, Maximum number of subjects = 1,000
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AKL-T01 (EVO Multi) (Active Comparator): AKL-T01, or EVO Multi, is a digital intervention that requires the subject to navigate a character through a game-like space, while collecting objects, in a fixed period of time.
  Interventions: Device: AKL-T01
- AKL-T09 (EVO Words) (Active Comparator): AKL-T09, or EVO Words, is a digital intervention that requires the subject to spell as many words as possible, by connecting letters in a game-like grid, in a fixed period of time.
  Interventions: Device: AKL-T09

INTERVENTIONS:
Device: AKL-T01 — Videogame-like digital therapy
  Other Names: EVO Multi
  Arms: AKL-T01 (EVO Multi)
Device: AKL-T09 — Videogame-like digital therapy
  Other Names: EVO Words
  Arms: AKL-T09 (EVO Words)

SUMMARY:
The purpose of this study is to evaluate the effects of videogame-like digital therapies on attentional functioning and symptoms in children diagnosed with ADHD.

DETAILED DESCRIPTION:
The study will be a randomized, parallel group, controlled trial of two videogame-like (iPad-based) digital therapies. The study will consist of 3 primary phases: Screening, Washout/Baseline, and Treatment. During the Screening Phase (Day -28 to Day -7), participants will undergo screening to evaluate eligibility for the study. Screening may take place up to 28 days before the Baseline Visit (Day 0). For those children currently on medication for ADHD the Washout period will begin 7 days prior to Baseline where treatment will be discontinued. On Day 0, the Baseline visit will occur wherein additional eligibility criteria will be established. The Treatment Phase (Day 1 to Day 27) will involve using the digital therapy at home for each participant followed by an In-Clinic assessment on Day 28 to assess key outcomes. Compliance with treatment/use requirements will be monitored remotely during this phase.

ELIGIBILITY:
Inclusion Criteria:

Confirmed ADHD diagnosis, any presentation, at Screening based on the Diagnostic and Statistical Manual of Mental Health-Fifth Edition criteria and established via the MINI-International Neuropsychiatric Interview for Children and Adolescents administered by a trained clinician

Screening/Baseline score on the clinician-rated ADHD-RS-IV score >= 28

Screening/Baseline score on the TOVA 8 API <= -1.8

Not undergoing pharmacological treatment with methylphenidate or amphetamine-based products at time of Screening; or, if undergoing pharmacological treatment, must be willing and appropriate (i.e. not optimally treated in the investigator's judgment) to wash out of current regimen

Ability to follow written and verbal instructions (English), as assessed by the PI

Estimated Intelligence Quotient score >= 80 as assessed by the Kaufmann Brief Intelligence Test, Second Edition (KBIT-II)

Ability to comply with all the testing and requirements.

Exclusion Criteria:

Current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis, based on MINI-KID and subsequent clinical interviewing, with significant symptoms including but not limited to post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator that may confound study data/assessments. Participants with clinical history of learning disorders will be allowed to participate, provided the disorder does not impact their ability to participate in the trial based on PI judgment

Participants who are currently treated with a non-stimulant medication for ADHD (i.e., atomoxetine, clonidine clonidine, guanfacine)

Initiation within the last 4 weeks of behavioral therapy. Participants who have been in behavior therapy consistently for more than 4 weeks may participate provided their routine is unchanged during the course of the study. Participants planning on changing or initiating behavior therapy during the course of the study will be excluded

Participant is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation or self-injurious behavior as measured by Columbia Suicide Severity Rating Scale at screening

Motor condition (e.g., physical deformity of the hands/arms; prostheses) that prevents game playing as reported by the parent or observed by the investigator

Recent history (within the past 6 months) of suspected substance abuse or dependence

History of seizures (exclusive of febrile seizures), or significant motor or vocal tics, including but not limited to Tourette's Disorder

Has participated in a clinical trial within 90 days prior to screening

Diagnosis of or parent-reported color blindness (Confirmed in-clinic via ICBT)

Uncorrected visual acuity (Confirmed in-clinic via ability of subject to play the intervention)

Regular use of psychoactive drugs (other than stimulant) that in the opinion of the Investigator may confound study data/assessments

Any other medical condition that in the opinion of the investigator may confound study data/assessments

Has a sibling also enrolled/currently participating in the same study

Has previously participated in a study of Akili's EVO videogame-like digital therapy

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kollins, PhD, Principal Investigator — Duke Clinical Research Institution
Locations (20):
- United States (20):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Melmed Center, Scottsdale, Arizona
  - Avida, Inc., Newport Beach, California
  - University of California Davis MIND Institute, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Meridien Research, Bradenton, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - South Shore Psychiatric Services, Marshfield, Massachusetts
  - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Duke Child and Family Study Center, Durham, North Carolina
  - The Neuropsychiatric Clinic at Carolina Partners, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - FutureSearch Trials, Dallas, Texas
  - Bayou City Research, Ltd, Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stamatis CA, Heusser AC, Simon TJ, Ala'ilima T, Kollins SH. Real-time cognitive performance metrics derived from a digital therapeutic for inattention predict ADHD-related clinical outcomes: Replication across three independent trials of AKL-T01. Transl Psychiatry. 2024 Aug 11;14(1):328. doi: 10.1038/s41398-024-03045-0. PMID 39128918
- [Derived] Kollins SH, DeLoss DJ, Canadas E, Lutz J, Findling RL, Keefe RSE, Epstein JN, Cutler AJ, Faraone SV. A novel digital intervention for actively reducing severity of paediatric ADHD (STARS-ADHD): a randomised controlled trial. Lancet Digit Health. 2020 Apr;2(4):e168-e178. doi: 10.1016/S2589-7500(20)30017-0. Epub 2020 Feb 24. PMID 33334505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met full criteria for ADHD at Screening and who the PI believed were not optimally treated with current medication were eligible to washout their medication regimen. For those electing to washout, treatment was discontinued between 7 and 3 days prior to their scheduled Baseline Visit.
Period: Overall Study
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Started | 180 | 168
Completed | 175 | 164
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words) | Total
Number analyzed (Participants) | 180 | 168 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.711 (1.322) | 9.601 (1.341) | 9.658 (1.331)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 45 | 100
  Male | 125 | 123 | 248
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 133 | 119 | 252
  Black or African American | 25 | 26 | 51
  Other | 22 | 23 | 45
Region of Enrollment [Number; unit: participants]
  United States | 180 | 168 | 348

OUTCOME MEASURES:

1. Primary Outcome: Test of Variables of Attention-Attention Performance Index (Change From Baseline to Posttreatment)
Description: TOVA API is a comparison of the subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. The API is calculated from variability, response time, and d' (D Prime) using the following formula:
  API = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80 where Response Time is the average time it takes to respond correctly to a target, d' score is a response discriminability score reflecting the ratio of hits to "false alarms", and Variability is a measure of consistency of speed of responding based on the standard deviation of the mean correct response times. API tells how similar the score is to the ADHD profile. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.
  The calculation for difference in TOVA API was API at Day 28 minus API at Day 0 of this study.
Time Frame: Day 0 to Day 28
Population: Intent to Treat Population - all randomized participants
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 180 | 168
z-score | 0.93 (3.2) | 0.03 (3.2)

2. Secondary Outcome: ADHD-RS Total (Change From Baseline to Posttreatment)
Description: The ADHD-RS-IV is an 18-item, clinician-administered questionnaire for which a parent respondent rates the frequency of occurrence of ADHD symptoms and behaviors as defined by criteria outlined for ADHD in the DSM-IV. Each item is scored on a 4-point scale ranging from 0 (rarely or never) to 3 (very often) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors. A negative change in total score indicates improvement from Day 0 to Day 28.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all randomized participants) from whom both Day 0 and Day 28 data was able to be collected in full. For the ADHD-RS, this population included all participants for whom all 18 items of the rating scale were completed. In the AKL-T01 arm, two participants were missing a response for at least one item of the ADHD-RS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 173 | 164
score on a scale | -6.2 (7.6) | -5.7 (8.2)

3. Secondary Outcome: ADHD-RS Inattentive Subscale (Change From Baseline to Posttreatment)
Description: The ADHD-RS-IV is an 18-item, clinician-administered questionnaire for which a parent respondent rates the frequency of occurrence of ADHD symptoms and behaviors as defined by criteria outlined for ADHD in the DSM-IV. Each item is scored on a 4-point scale ranging from 0 (rarely or never) to 3 (very often) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors.
  The 18 items are grouped into 2 subscales: hyperactivity/impulsivity (even numbered items 2-18) and inattentiveness (odd numbered items 1-17). Each subscale produces a sub-scale score ranging from 0-27. A higher subscale score indicates more severe ADHD symptoms and behaviors.
  A negative change indicated improvement on the subscale from Day 0 to Day 28.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all randomized participants) from whom both Day 0 and Day 28 data was able to be collected in full. For the ADHD-RS, this population included all participants for whom all 9 items of the sub-scale were completed. In the AKL-T01 arm, two participants were missing a response for at least one item of the sub-scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 173 | 164
score on a scale | -3.6 (4.8) | -3.2 (5.0)

4. Secondary Outcome: ADHD-RS Hyperactivity Subscale (Change From Baseline to Posttreatment)
Description: as for outcome 3
Time Frame: Study Day 0 to Study Day 28
Population: Intent to Treat Population - all randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 175 | 164
score on a scale | -2.6 (4.2) | -2.5 (4.5)

5. Secondary Outcome: BRIEF Working Memory Percentile (Change From Baseline to Posttreatment)
Description: The Behavior Rating Inventory of Executive Function (BRIEF) is a parent-rated form that assesses everyday behavior associated with specific domains of the executive functions of their child. The BRIEF working memory metacognition subscale measures the participants ability to hold information when completing a task in a sequential manner.
  A negative change in percentile indicated an improvement on the subscale.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT from whom both Day 0 and Day 28 data was able to be collected in full. For the BRIEF WM, this includes all participants for whom all items of the sub-scale were completed. In both the AKL-T01 and AKL-T09 arms 9 participants were missing a response for at least one item (18 total participants were missing responses to items).
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 166 | 155
percentile | -3.1 (8.0) | -3.3 (9.4)

6. Secondary Outcome: BRIEF Inhibit Percentile (Change From Baseline to Posttreatment)
Description: The Behavior Rating Inventory of Executive Function (BRIEF) is a parent-rated form that assesses everyday behavior associated with specific domains of the executive functions of their child. The BRIEF Inhibit subscale measures the participant's ability to control impulses and to stop engaging in a behavior.
  A negative change in percentile indicated an improvement on the subscale.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT from whom both Day 0 and Day 28 data was able to be collected in full. For BRIEF Inhibit this includes all participants for whom all items of the sub-scale were completed. In both the AKL-T01 and AKL-T09 arms 9 participants were missing a response for at least one item (18 total participants were missing responses to items).
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 166 | 155
percentile | -2.8 (13.3) | -3.5 (9.2)

7. Secondary Outcome: Impairment Rating Scale, Overall Impairment (Change From Baseline to Posttreatment)
Description: The Impairment Rating Scale (IRS) is a parent-rated scale that assesses individualized areas of impairment for a child participant and asks parents to make a rating of how significantly these problems impact functioning across a range of domains (social, family, school, self-esteem). Parents describe the primary areas of difficulty for each child and then provide a rating (via a Visual Analog Scale) of how much the difficulties affect the different areas of functioning ranging from (1) "no problem; definitely does not need treatment or special services" to (7) "extreme problem; definitely needs treatment or special services."
  The total IRS is 8 items, the 8th rating overall impairment. A negative change indicated a decrease in overall impairment.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT from whom both Day 0 and Day 28 data was able to be collected in full. For the IRS, this includes all participants for whom item #8 (overall impairmant) was completed. In the AKL-T01 arm, item #8 was not answered by 4 participants. In the AKL-T09 arm, item #8 was not answered by 3 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 171 | 161
score on a scale | -0.5 (1.4) | -0.4 (1.2)

8. Secondary Outcome: CGI-I (at Posttreatment)
Description: The Clinical Global Impression Scale - Improvement (CGI-I) is a clinician's comparison of the participant's overall clinical condition at follow up to the overall clinical condition at baseline. The CGI-S is a 7-point scale where 1 = Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse.
  A score of 1, 2, or 3 would indicate overall improvement of ADHD severity.
Time Frame: Day 28
Population: Intent to Treat Population - all randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 175 | 164
score on a scale | 3.4 (0.9) | 3.4 (0.9)

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/168
Other Adverse Events (participants affected / at risk) | 12/180 | 3/168
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKL-T01 (EVO Multi) (N=180) | AKL-T09 (EVO Words) (N=168)
Nausea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0
Frustration tolerance decreased (Psychiatric disorders) | 5 | 0
Emotional disorder (Psychiatric disorders) | 2 | 1 — The lower level term 'emotional reaction' better describes the verbatim term reported from the site.
Aggression (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02674633/Prot_SAP_000.pdf